CLINICAL TRIAL: NCT04519333
Title: Intradermal Mesotherapy Versus Systemic Therapy in Treating Neck Pain to Cervical Disc Herniation: A Prospective Randomized Study
Brief Title: Mesotherapy Versus Systemic Therapy in Treating Neck Pain Related to Herniated Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Principal Investigator, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AtaturkU0001
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Emergencies
Keywords: Mesotherapy; Neck Pain
MeSH Terms: conditions — Emergencies; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compare to sistemic treatment and mesotherapy. (Other): This is a prospective parallel randomized controlled trial conducted with patients admitted to our emergency department with neck pain related to cervical disc herniation
  Interventions: Procedure: drug(intradermal injection)

INTERVENTIONS:
Procedure: drug(intradermal injection) — The mesotherapy was performed by an experienced and trained physician using a disposable 4 mm and 6 mm long, 30 Gauge needles. Initially, a pharmacological mixture of 1 cc (2 mg) thiocolchicoside, 1 cc (16.2 mg) lidocaine and 1 cc (5 mg) tenoxicam was prepared for each treatment session, and 0.1-0.2 cc of this mixture was applied to each injection point with a depth of 1-3 mm using point by point intradermal method without causing papules.
  In the systemic therapy group, we applied a 50 mg dexketoprofen (Revafen, Haver Pharma Pharmaceutical Co., Turkey) in 100 cc isotonic solution intravenously for 5 minutes.

SUMMARY:
Introduction: Neck pain is a global public health concern, that ranked 4th highest health condition in terms of disability as measured by years lived with disability. The aim of this study is to compare the efficiency of one-session mesotherapy application with systemic therapy in treating neck pain related to cervical disk herniation.

Methods: This is a prospective parallel randomized controlled trial conducted with patients admitted to our emergency department with neck pain related to cervical disc herniation. A mixture of thiocolchicoside, lidocaine and tenoxicamwas administered via mesotherapy in one group, and intravenous administration of dexketoprofen was applied to the other group. We compared the changes in pain intensity at 60thminute, 120thminute and 24th hours after treatment using Visual Analogue Scale (VAS),and adverse effects of the treatment methods among the study groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older age
* Admission to Emergency Department (ED) with acute cervical pain related to cervical disk herniation.

Exclusion Criteria:

* Taking analgesic drugs before admission
* Having VAS score of lower than 4 on admission
* Having diabetes mellitus
* Body mass index>30 kg/m2
* Pregnancy
* Lactation
* Having active bleeding or bleeding disorder
* Having active or recurrent gastrointestinal hemorrhage or ulcer, or history of these conditions
* Having a serious or life-threatening condition (stroke, intracranial hemorrhage, heart attack, cardiac tamponade, pneumothorax, hemothorax, flail chest, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | 0-24 hours
  we defined as the delta value of Vizuel Analog Score(points between 0-10,the most severe pain 10 points,0 points no pain) scores with different time intervals. We calculated delta values by subtracting the VAS scores at 60th and 120th minutes, and 24th hours from the VAS score on admission.
Adverse effect | 0-1 week
  we have defined as the presence of hypotension, dizziness, nausea, vomiting, diarrhea, edema, localized infections, pruritus, bruising or swelling at the injection sites in the mesotherapy group; and presence of dry mouth, hypotension, dizziness, nausea, vomiting, diarrhea, dyspepsia, peptic ulceration, peptic ulcer bleeding, urticarial lesion, pruritus in the systemic therapy group. The patients were followed up for one week for presence of adverse effects. We interviewed with the patientsdaily by telephone for adverse effects, and evaluated all the patientswith an ED visit at the end of follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No